CLINICAL TRIAL: NCT00345592
Title: TReatment of Atrial Fibrillation With Dual dEfibrillator in Heart Failure Patients
Acronym: TRADE HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005_TH
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device managed arm (Experimental): Device-managed therapy arm. Shock therapy for atrial arrhythmias is delivered automatically from the device.
  Interventions: Device: Dual (atrial and ventricular) implantable defibrillator
- Traditional arm (Active Comparator): Traditional therapy arm. In this arm, therapy for atrial arrhythmias will be delivered from the device through command of the physician and in a hospital environment. Therefore, patients who will experience symptoms at home, will refer to their center, eventually hospitalized and treated for atrial arrhythmias.
  Interventions: Device: Dual (atrial and ventricular) implantable defibrillator

INTERVENTIONS:
Device: Dual (atrial and ventricular) implantable defibrillator — The devices automatically applies therapy (shock) for atrial fibrillation, when atrial fibrillation is confirmed.
  Arms: Device managed arm
Device: Dual (atrial and ventricular) implantable defibrillator — In hospital application of anti arrhythmic therapies via the device
  Arms: Traditional arm
Device: Dual (atrial and ventricular) implantable defibrillator — Therapy for atrial arrhythmias will be delivered from the device through command of the physician and in a hospital environment
  Arms: Traditional arm

SUMMARY:
Demonstrate the efficacy of the device-based managed therapy to treat atrial tachycardia and fibrillation (AT/AF) in patients with CHF indication for implant of a CRT defibrillator and to demonstrate the advantage of automatic electrical therapy of atrial arrhythmias compared to an in-hospital approach for treatment of symptomatic AT/AF.

ELIGIBILITY:
Inclusion Criteria:

* chronic symptomatic HF despite stable, optimal drug therapy
* indication for a cardiac resynchronisation device with defibrillator backup according to current guidelines
* patients implanted with cardiac resynchronization device with dual (atrial and ventricular) defibrillation capabilities

Exclusion Criteria:

* Chronic atrial fibrillation
* Valvular disease
* patients who underwent or are planned for ablation of atrial fibrillation
* cerebral vascular accident/transient ischemic attack within 12 months from implant which lead to relevant impairment
* preexisting unipolar pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2006-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Botto, MD, Principal Investigator — Azienda Ospedale S. Anna; Luigi Padeletti, MD, Principal Investigator — Istituto di Clinica Medica I° e Cardiologia A.O.C. Careggi
Locations (2):
- Italy (2):
  - Istituto di Clinica Medica I° e Cardiologia A.O.C., Careggi
  - Azienda Ospedale S. Anna, San Fermo Della Battaglia (CO)

REFERENCES:
- [Derived] Botto GL, Boriani G, Favale S, Landolina M, Molon G, Tondo C, Biffi M, Grandinetti G, De Filippo P, Raciti G, Padeletti L. Treatment of atrial fibrillation with a dual defibrillator in heart failure patients (TRADE HF): protocol for a randomized clinical trial. Trials. 2011 Feb 15;12:44. doi: 10.1186/1745-6215-12-44. PMID 21324118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on the 3rd of October, 2006. Last patient was enrolled on the 29th of July 2009, for a total of 420 patients.
Pre-assignment Details: 24 subjects were not randomized:
  * 7 died before randomization (causes: 3 cardiac, 2 non-cardiac, 2 unknown);
  * 7 voluntarily withdrew;
  * 5 withdrawn due to AF.
  * 2 had device explanted before randomization;
  * 1 had biventricular pacing turned OFF
  * 1 was withdrawn from the study for inclusion criteria violation;
  * 1 lost to follow up.
Period: Overall Study
Arm/Group | Device Managed Arm | Traditional Arm
Started | 199 | 197
Completed | 174 | 173
Not Completed | 25 | 24
Not completed — Death | 14 | 16
Not completed — Withdrawal by Subject | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Managed Arm | Traditional Arm | Total
Number analyzed (Participants) | 199 | 197 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 68 (10) | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 38 | 85
  Male | 152 | 159 | 311
Region of Enrollment [Number; unit: participants]
  Italy | 199 | 197 | 396

OUTCOME MEASURES:

1. Primary Outcome: Unplanned Hospital Admissions for Cardiac Reasons OR Death of Cardiovascular Causes OR Progression to Chronic Atrial Fibrillation
Time Frame: 3 years from randomization (39 months total)
Measure: Number; unit: participants
Arm/Group | Device Managed Arm | Traditional Arm
Number analyzed (Participants) | 199 | 197
participants | 43 | 44
Statistical Analysis 1: Comparison: Device Managed Arm vs Traditional Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.987, 95% CI 2-sided [0.684 to 1.503]

ADVERSE EVENTS:
Arm/Group | Device Managed Arm | Traditional Arm
Serious Adverse Events (participants affected / at risk) | 103/199 | 93/197
Other Adverse Events (participants affected / at risk) | 39/199 | 22/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Managed Arm (N=199) | Traditional Arm (N=197)
atrial fibrillation (Cardiac disorders) | 10 (11) | 7 (9)
worsening of cardiac disorders (Cardiac disorders) | 16 (16) | 14 (14) — events leading to death
hopspitalizatin/intervention (General disorders) | 78 (85) | 58 (74) — including cardiac and non cardiac hospitalizations
transplant (Cardiac disorders) | 6 (6) | 4 (4)
worsening of non-cardiac disorders (General disorders) | 8 (8) | 10 (10) — events leading to death
worsening of unknown conditions leading to death (General disorders) | 13 (13) | 7 (7) — include all the events leading to out of hospital death for unknown or undetermined conditions
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Managed Arm (N=199) | Traditional Arm (N=197)
device reprogramming (Cardiac disorders) | 16 (17) | 14 (15) — need to change device settings due to patient sysmptoms or adverse device effect, without invasive intervention
clinical observation (General disorders) | 24 (24) | 8 (8) — not requiring intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No